CLINICAL TRIAL: NCT03244904
Title: a Prospective Cohort Study for Small Cell Lung Cancer to Identify Susceptibility Gene and Assess DNA Dynamic Change by Next-generation Sequencing
Brief Title: Next-generation Sequencing of Small Cell Lung Cancer to Identify Susceptibility Gene and to Assess Treatment
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Fujian Cancer Hospital (Other Government)
Responsible Party: Sponsor
Other Study IDs: CSWOG01
Record Dates: First submitted 2017-08-05; First posted 2017-08-10 (Actual); Last update posted 2017-08-10 (Actual); Status verified 2017-07

CONDITIONS: SCLC
Keywords: NGS,SCLC, ctDNA

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective

SUMMARY:
Participants will be consented into the study after they are found to meet the study inclusion criteria. The clinical staff will schedule a tissue biopsy and a blood draw for the participant to give NGS(Next-generation Sequencing).One is according to the germline mutation data to screen susceptible gene in SCLC(Small Cell Lung Cancer); two is to explore the extensive consistency detection of blood and tissues in patients with SCLC gene mutation information; three is to conduct dynamic monitoring of blood ctDNA(circulating tumor DNA) in patients with SCLC during treatment, by changing the types of mutations / abundance (for example: the clonal evolution of typical samples analysis) and change of tumor load, , investigating the patients treatment effect , for the significant change of mutations, to study whether it can be used as molecular marker; four is to analyze of the molecular typing of SCLC, according to the clinical and pathological features of patients.

ELIGIBILITY:
Inclusion Criteria:

* Patients must understand the rigors of the study and provide written informed consent and HIPAA authorization prior to initiation of any study procedures
* Life expectancy > 10 months
* Karnofsky Performance Status ≥ 70
* Diagnosis of histological or cytologically confirmed SCLC,
* Age ≥ 18 years
* Good medical candidate for and willing to undergo a biopsy or surgical procedure to obtain tissue, which may or may not be part of the patient's routine care for their malignancy.

Exclusion Criteria:

* Poor compliance, reluctant to undergo research medication, or follow-up.
* Tumor inaccessible for biopsy
* It is currently included in clinical trials of other drugs, or at the same time, into other medical studies that are considered incompatible with the study.
* It has a history of other cancers, unless the cancer is completely relieved and has not been treated for more than 3 years.

Ages: 18 Years to 70 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: SCLC
Sampling Method: Non-Probability Sample
Enrollment: 80 (Estimated)
Dates: Start 2017-11 (Estimated); Primary Completion 2017-11 (Estimated); Study Completion 2018-07 (Estimated)

PRIMARY OUTCOMES:
susceptibility gene site of small cell lung cancer | 01.11.2017-31.05.2018
  searching susceptibility gene site of small cell lung cancer according to germline mutation data

SECONDARY OUTCOMES:
consistency of ctDNA and tDNA sequencing results in patients with SCLC | 01.11.2017-31.05.2018
  explore consistency of ctDNA and tDNA sequencing results in patients with ESCLC

OTHER OUTCOMES:
sensitive molecular markers for treating | 01.11.2017-31.05.2018
  during treatment of blood ctDNA for dynamic monitoring, through the mutation type/abundance changes (for example, a typical sample of clonal evolution analysis) and tumor mutation load change, studying whether significant changes of mutations can be used as molecular markers of SCLC
molecular classification of SCLC | 01.11.2017-31.05.2018
  according to the clinicopathological features of the patients with sclc enrolled , analyzeing molecular classification of SCLC by analyzing mutation types

CONTACTS AND LOCATIONS:
Overall Officials: Gen Lin, MD,PhD, Principal Investigator — CSWOG

IPD SHARING:
Plan to Share IPD: Undecided